CLINICAL TRIAL: NCT02413086
Title: Effectiveness and Safety of Early-Stage Amputation and External Herbs Chitosan for Diabetic Foot Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wang Kuanyu, Director of Department of Surgery, First Affiliated Hospital of Heilongjiang UCM, Heilongjiang University of Chinese Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ESA-EHC-DFU-2014
Record Dates: First submitted 2015-03-23; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetic foot ulcer; early-stage amputation; external therapy of herbs chitosan; wound surface healing
MeSH Terms: conditions — Diabetic Foot | interventions — Amputation, Surgical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Early-stage amputation+external herbs chitosan (Experimental): Individuals with DFU were given early-stage amputation and wound was given herbs chitosan after amputation.
  Interventions: Procedure: Early-stage amputation; Other: External herbs chitosan
- Early-stage amputation+traditional gauze (Experimental): Individuals with DFU were given early-stage amputation and wound was given traditional gauze after amputation.
  Interventions: Procedure: Early-stage amputation; Other: Traditional gauze
- Amputation+external herbs chitosan (Experimental): Individuals with DFU were given amputation and wound was given herbs chitosan after amputation.
  Interventions: Procedure: Amputation; Other: External herbs chitosan
- Amputation+traditional gauze (Experimental): Individuals with DFU were given amputation and wound was given traditional gauze after amputation.
  Interventions: Procedure: Amputation; Other: Traditional gauze

INTERVENTIONS:
Procedure: Early-stage amputation — Individuals with DFU were given early-stage amputation.
  Arms: Early-stage amputation+external herbs chitosan; Early-stage amputation+traditional gauze
Procedure: Amputation — Individuals with DFU were given amputation.
  Arms: Amputation+external herbs chitosan; Amputation+traditional gauze
Other: External herbs chitosan — Wound was given external herbs chitosan after amputation.
  Arms: Amputation+external herbs chitosan; Early-stage amputation+external herbs chitosan
Other: Traditional gauze — Wound was given traditional gauze after amputation.
  Arms: Amputation+traditional gauze; Early-stage amputation+traditional gauze

SUMMARY:
Diabetic Foot as the popular chronic complications of diabetes, is one of the main factors leading to limb amputation, it was reported that the amputation rate is 15 times of the non-diabetic patients. Common surgical amputation is not only about high plane amputation but also bring a tremendous mental stress to patients which may affect the quality of life seriously. Diabetic foot patients facing the great risk of serious infection, endotoxemia , and septic shock which could be the main cause of death before amputation. It become an important topic that how to control the infection, reduce the amputation plane, save the function as possibility, and improve the life quality of the patients as well.

This study is based on years of clinical experience of and brings out "early-stage amputation" concept firstly in China with a systematic exposition, experimental research and clinical research. Early-stage amputation refers to cut in the normal tissue from the inflammatory tissue at the junction line of limbs, in order to achieve more retained stump, block endotoxin absorption and improve the quality of life of patients. External therapy of herbs chitosan can promote granulation tissue regeneration and control of local infection, it solved the problem of difficult wound healing and it is a reliable guarantee of early-stage amputation.

ELIGIBILITY:
Inclusion Criteria:

1. According to Chinese herbs medicine standard for the diagnosis and treatment of diabetic foot, the individual diagnosed as diabetic foot with acromelic gangrene.
2. The individual aged between 18 and 70 years.
3. All wounds corresponded to Wagner classification grade 4 or 5.
4. By appropriate treatment, skin temperature of limb with ulcer became warmer and it proved that the blood circulation recovery could be happening.
5. There were no obvious bruises or chromatosis in the necrosis skin.
6. Persistent limb pain affected the sleep of the individuals.
7. The individual voluntarily signed the informed consent form.

Exclusion Criteria:

1. Acromelic gangrene caused by other reasons.
2. The individuals with server cardiovascular and cerebrovascular diseases or hepatic and kidney diseases do not adhere to surgery.
3. The individuals with the history of amputation.
4. The individuals with systemic inflammatory response syndrome, Bacteremia, Pyemia or shock.
5. Vascular ultrasound shows artery is completely blocked.
6. The individuals do not adhere to the treatment or are with other treatments.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The re-operation rate | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
  Because of diabetic foot ulcer individual was given a re-operation.
Grades of wound healing | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
  As wound healing, wound healing was assessed using 1 to 3 healing grades.

SECONDARY OUTCOMES:
Healing time | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
  After amputation the time to heal.
The rate of infection | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.
  After amputation, there was infection or no infection in the wound.
Amputation level | At time of surgery.
  Amputation level includes metatarsophalangeal joint, metatarsus, foot, ankle, below knee and the lower part of the thigh.
Trinity amputation and prosthesis experience scale (TAPES) | 7 days of amputation, 14 days of amputation, 1 month of amputation, 3 months of amputation and 6 months of amputation.
SF-36 | 7 days of amputation, 14 days of amputation, 1 month of amputation, 3 months of amputation and 6 months of amputation.
  The medical outcomes study 36-item short form health survey

CONTACTS AND LOCATIONS:
Overall Officials: Wang Kuang Yu, Doctor, Principal Investigator — First Affiliated Hospital of Heilongjiang UCM

REFERENCES:
- [Result] Armstrong DG, Lavery LA; Diabetic Foot Study Consortium. Negative pressure wound therapy after partial diabetic foot amputation: a multicentre, randomised controlled trial. Lancet. 2005 Nov 12;366(9498):1704-10. doi: 10.1016/S0140-6736(05)67695-7. PMID 16291063
- [Result] Jiang Y, Ran X, Jia L, Yang C, Wang P, Ma J, Chen B, Yu Y, Feng B, Chen L, Yin H, Cheng Z, Yan Z, Yang Y, Liu F, Xu Z. Epidemiology of type 2 diabetic foot problems and predictive factors for amputation in China. Int J Low Extrem Wounds. 2015 Mar;14(1):19-27. doi: 10.1177/1534734614564867. Epub 2015 Jan 8. PMID 25573978
- [Result] Yang SH, Dou KF, Song WJ. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Jun 24;362(25):2425-6; author reply 2426. No abstract available. PMID 20578276
- [Result] Collier A, Dowie A, Ghosh S, Brown PC, Malik I, Boom S. Diabetic foot ulcer: amputation on request? Diabetes Care. 2011 Oct;34(10):e159. doi: 10.2337/dc10-2183. No abstract available. PMID 21949231
- [Result] Attinger C, Venturi M, Kim K, Ribiero C. Maximizing length and optimizing biomechanics in foot amputations by avoiding cookbook recipes for amputation. Semin Vasc Surg. 2003 Mar;16(1):44-66. doi: 10.1053/svas.2003.50006. No abstract available. PMID 12644975